CLINICAL TRIAL: NCT05039892
Title: An Open-label, Single Arm, Multicenter Phase 2 Study to Evaluate the Efficacy and Safety of 3D185 Monotherapy in Subjects With Previously Treated Locally Advanced or Metastatic Cholangiocarcinoma With FGFR2 Gene Alterations
Brief Title: Efficacy and Safety of 3D185 Monotherapy in Subjects With Previously Treated Locally Advanced or Metastatic Cholangiocarcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: 3D Medicines (Beijing) Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: 3D Medicines (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3D185-C-002
Record Dates: First submitted 2021-09-02; First posted 2021-09-10 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Cholangiocarcinoma,Adult
MeSH Terms: conditions — Cholangiocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- All eligible subjects (Experimental)
  Interventions: Drug: 3D185

INTERVENTIONS:
Drug: 3D185 — All eligible subjects will receive the RP2D regimen to be established based on the results of the ongoing phase I study from Cycle 1 Day 1 (C1D1) until disease progression, intolerable toxicity, withdrawal of consent, whichever occurs first.

SUMMARY:
The purpose of this study is evaluate the efficacy of 3D185 in subjects with advanced/metastatic cholangiocarcinoma with FGFR2 Gene Alterations who have failed at least 1 previous treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed cholangiocarcinoma.
2. Documented disease progression following at least one previous systemic cancer therapy
3. Tumor assessment for FGF/FGFR gene alteration status.
4. Have measurable disease according to RECIST v1.1
5. ECOG Performance Status ≤ 2
6. Life expectancy ≥ 12 weeks.

Exclusion Criteria:

1. Previously received selective FGFR inhibitor therapy.
2. History of and/or current evidence of ectopic mineralization/calcification, including but not limited to soft tissue, kidneys, intestine, myocardia, or lung, excepting calcified lymph nodes and asymptomatic arterial or cartilage/tendon calcifications.
3. Have any of the following eye diseases/conditions: 1) history of retinal pigment epithelial detachment (RPED); 2) history of laser treatment or intraocular injection for macular degeneration; 3) history of dry or wet age-related macular degeneration; 4) history of retinal vein occlusion (RVO); 5) history of retinal degenerative diseases; 6) history of chorioretinal lesions..
4. Received CYP3A4 and/or CYP2C8 strong inhibitors or CYP3A4 strong inducers within 14 days prior to the first dose and subject who need to continue using these drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-12 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
ORR | 24 months
  defined as the proportion of subjects who achieved a confirmed complete response (CR) or partial response (PR) based on RECIST v1.1 as assessed by investigators.

SECONDARY OUTCOMES:
Duration of response (DoR) | 24 months
  DoR is defined as the time from the date of first CR or PR based on RECIST v1.1 to the date of first documented progressive disease based on RECIST v1.1 or death, whichever occurs first.
Disease control rate (DCR) | 24 months
  defined as the proportion of subjects who achieve a confirmed complete response (CR) or partial response (PR) or stable disease (SD) based on RECIST v1.1 as assessed by investigators.
Progression-free survival (PFS) | 24 months
  PFS is defined as the time from the date of first study dose to disease progression based on RECIST v1.1 or death, whichever occurs first.
Overall survival (OS) | 24 months
  OS is defined as the date of first study dose to the date of death from any cause.
3D185 Plasma concentration | 24 months
  The pharmacokinetic and pharmacodynamics assessments will be analyzed descriptively and presented in appropriate tables or figures.
Serum phosphate levels | 24 months
  The pharmacokinetic and pharmacodynamics assessments will be analyzed descriptively and presented in appropriate tables or figures.